CLINICAL TRIAL: NCT07257458
Title: Application of Methylation Markers in Early Detection and MRD Monitoring of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Yuqing Huang, Director, Beijing Haidian Hospital
Other Study IDs: M202535
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (NSCLC)
Keywords: cfDNA; Methylation biomarker; SHOX2; PTGER4; Surgery; MRD monitoring; Prognostic monitoring
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical treatment group: Patients treated with conventional surgical operations

SUMMARY:
This study aims to evaluate the utility of combined plasma SHOX2 and PTGER4 gene methylation analysis as a dynamic biomarker for monitoring minimal residual disease (MRD) and predicting recurrence in postoperative non-small cell lung cancer (NSCLC) patients. The primary objective is to determine whether serial methylation assessment can guide personalized adjuvant therapy decisions by identifying high-risk individuals, thereby potentially reducing overtreatment or undertreatment.

Stage I-IV NSCLC patients undergoing surgical resection were enrolled. Peripheral blood was collected longitudinally for circulating tumor DNA (ctDNA) methylation testing: preoperatively, postoperatively at 3 days, 1, 3, 6, 9, 12, 18, and 24 months, and upon radiographic recurrence. The dynamic changes in SHOX2/PTGER4 methylation levels and conventional tumor marker positivity rates were analyzed.

Comprehensive statistical analyses were performed: Correlation between methylation levels and radiographic findings was assessed using Pearson/Spearman tests; predictive accuracy for recurrence was evaluated via ROC curve analysis; patients were stratified into methylation-based risk groups; survival differences were compared using Kaplan-Meier curves with log-rank testing; independent predictive value was determined through multivariate Cox regression adjusting for clinicopathological confounders. Final efficacy assessment integrated ctDNA positivity timing, disease-free survival (DFS), and overall survival (OS) metrics.

This prospective biomarker study seeks to validate a novel epigenetic approach for postoperative management, potentially establishing ctDNA methylation monitoring as a standardized tool for MRD detection and recurrence risk stratification in resected NSCLC.

DETAILED DESCRIPTION:
Lung cancer has the highest global incidence and mortality among all malignancies. As a high-incidence country, China reported approximately 1.0606 million new cases and 733,300 deaths in 2022, accounting for 22.0% and 28.5% of all malignant tumors, respectively. While early surgery is the primary curative approach, the risk of postoperative recurrence is substantial, with 5-year recurrence rates of 19% for stage IA, 30% for stage IB, and 48.6% for stage II NSCLC. The 3-year recurrence rate for stage III patients is as high as 52%. Crucially, even when imaging confirms a "tumor-free status" (R0 resection), hidden minimal residual disease (MRD) often leads to recurrence.

Current MRD detection primarily analyzes mutations in circulating tumor DNA (ctDNA). However, high inter-patient mutational heterogeneity poses challenges for designing compact, broadly effective detection panels. The Tumor-informed approach, which designs patient-specific panels, is limited by its dependency on tumor tissue samples. In contrast, DNA methylation biomarkers for MRD analysis do not require prior knowledge of tumor-specific mutations. Their sensitivity is independent of high-frequency mutation burden, changes occur early in tumorigenesis, and they exhibit tissue and cancer type specificity. Furthermore, DNA methylation shows consistency across numerous genomic regions, enabling detection via multiple CpG sites.

The "Expert Consensus on Tumor DNA Methylation Biomarker Testing and Clinical Application (April 2024)" states that variations in DNA methylation levels are closely associated with tumor prognosis and can be used for MRD assessment and recurrence monitoring. Mounting evidence supports this: A 2023 BMC Medicine study of 195 NSCLC patients found that individualized methylation-based MRD monitoring signaled recurrence earlier than mutation-based monitoring. A 2023 JAMA Oncology study demonstrated that detecting ctDNA methylation of five genes could predict colorectal cancer recurrence up to 20 months earlier than imaging, with significantly higher recurrence risk in patients positive for ctDNA one month post-surgery (HR=17.5). Another prospective study (NCT00958737) in 805 colorectal cancer patients confirmed a significantly higher 2-year disease-free survival rate in the ctDNA methylation-negative group (82% vs 64%).

This study aims to investigate the role of plasma SHOX2 and PTGER4 gene methylation levels in monitoring MRD and evaluating efficacy in NSCLC patients post-surgery. The study will enroll patients with histopathologically/clinically diagnosed stage I-IV NSCLC undergoing surgical resection. Peripheral blood will be collected at multiple timepoints: pre-treatment, and post-treatment at 3 days, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, and upon recurrence for ctDNA methylation analysis.

Statistical analyses will include: Assessing the correlation between methylation levels and radiological metrics using Pearson or Spearman coefficients; Evaluating the predictive power for recurrence using Receiver Operating Characteristic (ROC) curves; Stratifying patients into high-risk and low-risk groups based on methylation results; Plotting recurrence-free survival curves using the Kaplan-Meier method and comparing groups with the Log-rank test; Assessing the independent predictive value of SHOX2 and PTGER4 methylation for recurrence risk using multivariate Cox regression analysis, adjusting for confounders like age, gender, and tumor stage; Finally, evaluating individualized therapeutic efficacy based on the timing of ctDNA positivity, Disease-Free Survival (DFS), and Overall Survival (OS). The goal is to provide a scientific basis for predicting recurrence risk and guiding treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-small cell lung cancer (NSCLC) by histopathology/clinical diagnosis.
* Age 18-85 years old.
* Lung cancer patients who are determined by clinicians to be eligible for surgical treatment.
* ECOG score ≤ 2, with an expected survival period of ≥ 6 months, and having signed the informed consent form.
* The subjects should have clear case information, including age, gender, and clinical diagnosis, etc.

Exclusion Criteria:

* Patients with a history of other malignant tumors or autoimmune diseases.
* Those with severe heart, lung or vascular diseases that make them unable to tolerate surgery.
* Pregnant or lactating women.
* Patients who may be unable to complete follow-up during the study, as well as other factors that the researcher deems inappropriate for participation in the study.
* Incomplete clinical or follow-up information.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer (NSCLC) diagnosed by histopathology/ clinical diagnosis and scheduled for surgical treatment were selected, with ages ranging from 18 to 85 years old. All enrolled patients had peripheral blood drawn within one week before treatment, and at 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months after treatment for the detection of SHOX2/PTGER4 methylation in plasma cell-free DNA DNA (cfDNA)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The median lead time of SHOX2/PTGER4 methylation compared with traditional methods (tumor markers, imaging) for prediction. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: SHOX2/PTGER4 Methylation Detection Kit (PCR Fluorescence Method).
Disease-free survival: Differences in DFS based on methylation status after treatment. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: Kaplan-Meier method.
Dynamic concentration changes: The relative change rate of methylation levels before and after treatment and during recurrence. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: SHOX2/PTGER4 Methylation Detection Kit (PCR Fluorescence Method).

SECONDARY OUTCOMES:
The rate of methylation "turning negative" after treatment | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: SHOX2/PTGER4 Methylation Detection Kit (PCR Fluorescence Method).
The relationship between methylation status and overall survival. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: Multivariate Cox regression, Log-rank test.
Forecast performance | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: Receiver Operating Characteristic Curve.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Huang, Principal Investigator — Beijing Haidian Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No